CLINICAL TRIAL: NCT00286767
Title: A Cohort Observational Study Evaluating Predictors, Incidence and Immunopathogenesis of Immune Reconstitution Syndrome (IRIS) in HIV-1 Infected Patients With CD4 Count Less Than or Equal to 100 Cells/microL Who Are Initiating Antiretroviral Therapy
Brief Title: Immune Reconstitution Syndrome in HIV-Infected Patients Taking Antiretroviral Therapy
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060086; 06-I-0086
Record Dates: First submitted 2006-02-03; First posted 2006-02-03 (Estimated); Last update posted 2019-10-07 (Actual); Status verified 2018-11-01

CONDITIONS: Immune Reconstitution Inflammatory Syndrome
Keywords: Opportunistic Infections; Immune Restoration Disease; Mycobacterial Infections; HIV-1 Infection; HIV; ART Naive
MeSH Terms: conditions — Immune Reconstitution Inflammatory Syndrome; Opportunistic Infections; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will investigate what factors may lead to the development of immune reconstitution syndrome (IRIS) in HIV-infected patients and what the outcome is after IRIS. It will also seek to better define and describe the syndrome. IRIS is a condition that can occur in HIV-infected people following the start of antiretroviral therapy. The sudden improvement of immune function with this therapy can cause an unexpected worsening of diseases the patient already has, such as tuberculosis or fungal infections, and development of fever, enlarged lymph nodes or other complications, or even uncover a previously silent disease.

HIV-infected people who are at least 18 years old, whose CD4+T cell count is 100 cells per microliter or less, and who have not previously been treated with combination antiretroviral therapy or have taken the drugs for less than 3 months and more than 6 months before screening for this study may be eligible to participate. Candindates must also live within the wider DC area so that acute problems after therapy initiation will be evaluated at NIH. Candidates are evaluated before starting therapy with a medical history and physical examination, blood and urine tests, electrocardiogram, chest x-ray and CT scan of the chest, tuberculin skin testing, apheresis, and possibly an intestinal (gut) and lymph node biopsy (surgical removal of a small piece of tissue for microscopic examination). For apheresis, blood is collected through a needle in an arm vein and spun in a machine that separates the blood components. The white blood cells and plasma are removed, and the red cells and platelets are returned through the same needle or through a needle in a vein in the other arm.

Participants have a complete history and physical examination and additional blood tests, including genetic studies, upon entering the study. They start taking anti-HIV medications, prescribed according to the current standard of care, as well as medications to treat other infections, and treatment of IRIS, if needed. The study lasts about 4 years. Patients return to the clinic at 2, 4, 8 and 12 weeks after the entry visit, then every 12 weeks (about every 3 months) until week 48 (the first year), and then every 16 weeks (about every 4 months) until the end of the study. At most visits, patients have a medical history, physical examination and blood and urine tests, including CD4+T cell count and HIV plasma viral load measurement. Apheresis is also done at weeks 24 and 48 and then once every 48 weeks. Intestinal and lymph node biopsies (optional) are also done at weeks 24 and 48. A syphilis test and PAP smear (for women) are done yearly. and plasma, cells and serum are stored at almost every visit for immunologic studies.

DETAILED DESCRIPTION:
A cohort observational study evaluating the predictors, incidence, clinical presentation and immunopathogenesis of Immune Reconstitution Syndrome (IRIS) in human immunodeficiency virus (HIV-1) infected patients with CD4 Count less than or equal to 100 cells/microL who are initiating antiretroviral therapy.

Immune reconstitution syndrome (IRIS) is a clinical syndrome that has been described in HIV infected patients after initiation of highly active anti-retroviral therapy (HAART), and is characterized by paradoxical acute worsening of an underlying opportunistic infection or AIDS-defining illness. There is no widely accepted syndromic definition, the pathogenesis of the syndrome is unclear and there is no specific therapy. The syndrome is more common in patients with low CD4+ T cell counts (less than 50 cells/microL) and in those with certain underlying infections (e.g. mycobacterial or cryptococcal infection) and is typically observed when there is evidence of response to HAART and while patients are still at risk for other opportunistic infections (OIs) or AIDS defining illnesses (e.g. pneumocystis jirovecii pneumonia or cytomegalovirus [CMV] retinitis). The incidence of IRIS varies depending on the studied population and is very frequent in developing countries creating significant diagnostic and therapeutic challenges as well as utilization of limited health resources.

DESIGN: International observational cohort study. Participants will be evaluated at baseline and followed according to the protocol follow up schedule after initiation of antiretroviral therapy for a total of two years. Acute symptoms that may be representing manifestations of IRIS will also be evaluated at additional acute care visits if necessary.

DURATION: Enrollment is ongoing. Each volunteer will be followed for at least two years. Total duration of the study will be approximately 8 years (including the optional extension phase in US).

SAMPLE SIZE: Approximately 600 patients will be enrolled, 200 in Kenya, 100 in Thailand and 300 in US. (enrollment is US will continue until approximately the other sites are full). Based on the incidence of IRIS in patients with low CD4 counts (approximately 20-40 percent), we anticipate strong power (approximately 90 percent) to identify baseline factors predictive of IRIS.

POPULATION: HIV-l-infected men and women, age greater than or equal to 18 years, antiretroviral therapy (ART)-naive with CD4+ T cell counts less than or equal to 100 cells/mm(3). Participants will be recruited and followed at three sites: the broader Washington DC, Kericho, Kenya and Bangkok, Thailand areas.

REGIMEN: Participants will be initiated on ART according to the clinical standard of care. If an OI or other AIDS defining illness is identified prior to or during screening or at any point during the study, they will also be treated according to standard of care.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. For the National Institutes of Health (NIH)/US site: HIV-1 infection, as documented by OraQuick rapid test using venipuncture whole blood, or fingerstick whole blood done at screening; or by reactive enzyme-linked immunosorbent assay (ELISA) and Western Blot as determined by NIH Clinical Pathology Laboratory or Leidos Biomedical Research, Inc. Monitoring Laboratory. HIV infection as determined by an outside Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory facility" will be accepted for enrollment and verified by a standard HIV-1 ELISA with Western Blot at NIH.

     For Keny Medical Research Institute/Walter Reed Project Clinical Research Center (KEMRI/WRP CRC)/Kenya site: HIV-1 infection will initially be diagnosed based upon two, serial rapid HIV tests according to Kenya Ministry of Health (MOH) guidelines. Volunteers entering this study will have HIV infection confirmed by two serial rapid HIV test in accordance with Kenya MOH guidelines and testing algorithm followed by a confirmation with a Western Blot using FDA approved-kits. Samples from participants with discrepant results (between the results from other institution and KEMRI/WRP-CRC laboratory) and/or indeterminate/negative Western Blot will be subjected to a nucleic acid assay i.e. DNA or RNA PCR. For Thailand, HIV-1 screening and confirmatory testing will be based on 3, HIV tests according to the Thai Ministry of Public Health guidelines. The subjects will initially be tested with a chemiluminescent microparticle immunoassay (CMIA) method that detects both HIV antigen and antibody. Confirmatory testing of HIV reactive samples by two different antibody detection methods will follow. Positive results by all three methods confirm HIV diagnosis. Discrepancy between the tests will require a nucleic acid detection method to confirm HIV diagnosis.
  2. No previous treatment with potent combination anti-retroviral therapy (ART), defined as any protease inhibitor (PI)-based or non-nucleoside reverse transcriptase inhibitor (NNRTI)-based regimen, or even triple nucleoside reverse transcriptase inhibitors (NRTI)-based regimen, consisting of at least three antiretroviral drugs (including a boosted PI with NNRTI combination). Patients with limited use of ART (less than 12 weeks duration) more than 24 weeks before screening will be eligible for study participation.
  3. Screening CD4+ cell count less than or equal to 100 cells/mm(3). * Note: CD4 < 100 cells/microL from an outside or the site s laboratory within 8 weeks prior to screening can be accepted as the screening value.
  4. Residence within the wider Washington D.C. area (approximately within a 120-mile radius from the NIH Bethesda campus) for the National Institutes of Health/US site and residents of the Kericho District Hospital catchment area, an approximate 93-mile (150 kilometers) radius, for the KEMRI/WRP CRC/Kenya site. Residence within the Bangkok Metropolitan area and nearby provinces are allowed to participate (approximately 120-mile radius from each of the clinical sites)
  5. Men and women age greater than or equal to 18 years.
  6. Ability and willingness of subject or legal guardian/representative to understand study requirements and give informed consent.
  7. Be willing to allow storage of blood or tissue samples for future research. (For Thailand: storage of blood or tissue samples is an optional procedure and therefore not a inclusion criteria)
  8. Be willing to have HLA testing. (For Thailand: HLA testing is an optional procedure and therefore not an inclusion criteria)
  9. For the NIH/US site: Participants should have a primary care physician or will need to agree to find one during the first 24-48 weeks on study. For the KEMRI/WRP/Kenya site: Participants must be enrolled in the Kericho District Hospital HIV Clinic. For the two Thailand clinical sites: participants must be enrolled in the HIV clinic at either of the sites.

EXCLUSION CRITERIA:

1. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
2. Pregnancy will be an exclusion criterion for study entry given the intense nature of the protocol regarding blood draws, diagnostic testing, and follow-up.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2006-02-01; Study Completion 2018-11-01

PRIMARY OUTCOMES:
To identify baseline predictors of IRIS within 6 months of HAART initiation prospectively in a group of HIV-1 infected patients with advanced disease who are starting antiretroviral therapy. | During the data analysis phase at the end of the study
To evaluate the immunopathogenesis of IRIS with the goal to identify more appropriate targets for future therapeutic interventions. | During the data analysis phase at the end of the study

SECONDARY OUTCOMES:
Evaluate the baseline clinical and immunological characteristics ofindividuals who develop IRIS and compare them with those who do not. | During the data analysis phase at the end of the study
To study the incidence and clinical manifestations of IRIS prospectively in a group of HIV-1 infected patients with advanced disease who are initiating antiretroviral therapy. | During the data analysis phase at the end of the study
To evaluate the impact of IRIS on the risk of subsequent death (attributable mortality). | During the data analysis phase at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Thailand (2):
  - The Thai Red Cross AID Research Center (TRC-ARC), Bangkok
  - Bamrasnaradura Infectious Disease Institute (BIDI), Nonthaburi

REFERENCES:
- [Background] French MA, Price P, Stone SF. Immune restoration disease after antiretroviral therapy. AIDS. 2004 Aug 20;18(12):1615-27. doi: 10.1097/01.aids.0000131375.21070.06. PMID 15280772
- [Background] French MA. Antiretroviral therapy. Immune restoration disease in HIV-infected patients on HAART. AIDS Read. 1999 Nov;9(8):548-9, 554-5, 559-62. PMID 11082733
- [Background] Shelburne SA, Visnegarwala F, Darcourt J, Graviss EA, Giordano TP, White AC Jr, Hamill RJ. Incidence and risk factors for immune reconstitution inflammatory syndrome during highly active antiretroviral therapy. AIDS. 2005 Mar 4;19(4):399-406. doi: 10.1097/01.aids.0000161769.06158.8a. PMID 15750393
- [Derived] Rocco JM, Laidlaw E, Galindo F, Anderson M, Sortino O, Kuriakose S, Lisco A, Manion M, Sereti I. Mycobacterial Immune Reconstitution Inflammatory Syndrome in HIV is Associated With Protein-Altering Variants in Hemophagocytic Lymphohistiocytosis-Related Genes. J Infect Dis. 2023 Jul 14;228(2):111-115. doi: 10.1093/infdis/jiad059. PMID 37040388
- [Derived] Vinhaes CL, Sheikh V, Oliveira-de-Souza D, Wang J, Rupert A, Roby G, Arriaga MB, Fukutani KF, Sawe F, Shaffer D, Ananworanich J, Phanuphak N, Andrade BB, Sereti I. An Inflammatory Composite Score Predicts Mycobacterial Immune Reconstitution Inflammatory Syndrome in People with Advanced HIV: A Prospective International Cohort Study. J Infect Dis. 2021 Apr 8;223(7):1275-1283. doi: 10.1093/infdis/jiaa484. PMID 32761193
- [Derived] Gouel-Cheron A, Nason M, Rupert A, Sheikh V, Robby G, Fahle GA, Sereti I. Cardiovascular Biomarker Profile on Antiretroviral Therapy Is Not Influenced by History of an IRIS Event in People With HIV and Suppressed Viremia. Open Forum Infect Dis. 2020 Jan 11;7(1):ofaa017. doi: 10.1093/ofid/ofaa017. eCollection 2020 Jan. PMID 32016127
- [Derived] Mahnke YD, Greenwald JH, DerSimonian R, Roby G, Antonelli LR, Sher A, Roederer M, Sereti I. Selective expansion of polyfunctional pathogen-specific CD4(+) T cells in HIV-1-infected patients with immune reconstitution inflammatory syndrome. Blood. 2012 Mar 29;119(13):3105-12. doi: 10.1182/blood-2011-09-380840. Epub 2012 Jan 4. PMID 22219223
- [Derived] Antonelli LR, Mahnke Y, Hodge JN, Porter BO, Barber DL, DerSimonian R, Greenwald JH, Roby G, Mican J, Sher A, Roederer M, Sereti I. Elevated frequencies of highly activated CD4+ T cells in HIV+ patients developing immune reconstitution inflammatory syndrome. Blood. 2010 Nov 11;116(19):3818-27. doi: 10.1182/blood-2010-05-285080. Epub 2010 Jul 26. PMID 20660788